CLINICAL TRIAL: NCT06880406
Title: Early Alterations of Peripheral Mitochondrial Function and Metabolomic Profile in Patients With Alzheimer's Disease and Related Dementias
Brief Title: Mitochondrial Function and Metabolomic Profile in Alzheimer's Disease and Related Dementias
Acronym: AMPAlz
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24-PP-19
Record Dates: First submitted 2025-03-07; First posted 2025-03-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; mitochondrial function; metabolomic
MeSH Terms: conditions — Alzheimer Disease | interventions — Mental Status and Dementia Tests; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALZHEIMER PATIENTS and NON ALZHEIMER PATIENTS (Experimental): Recruitment of 75 patients with amyloid positive marker on cerebrospinal fluid and 75 patients with amyloid negative marker on cerebrospinal fluid
  Interventions: Other: MMSE and blood draw

INTERVENTIONS:
Other: MMSE and blood draw — Each patient will be evaluated by Mini-Mental State Examination (MMSE) and will have a blood draw

SUMMARY:
This project aims to study on one hand the early mitochondrial alterations, common or specific, occurring in peripheral cells of patients with Alzheimer's disease or related dementia and, on the other hand, identify the metabolomic biomarkers that may be at the origin of mitochondrial disturbances associated with the disease. This will be the first study combining functional analyses of mitochondria and exploratory metabolomic assessments in the same cohort at early stages of the disease.

DETAILED DESCRIPTION:
Study will be proposed to the patient of the Nice Memory center who had a lumbar puncture and who agreed on the storage of a sample of their cerebrospinal fluid.

Two groups of patients will be compared: the Alzheimer"s disease patient with positive amyloid on the cerebrospinal fluid and the non Alzheimer patient with negative amyloid on the cerebrospinal fluid.

Blood samples will be collected at inclusion and one year to obtain the mitochondrial metabolomic signature

ELIGIBILITY:
Inclusion Criteria:

* Neurocognitive disorder with spontaneous complaint or reported for at least 6 months
* Diagnostic process according to current Haute Autorité de Santé (HAS) recommendations.
* cerebrospinal fluid biomarker dosage done within the study center and agreement to bio-collection of residual cerebrospinal fluid
* Patient having agreed to sign the informed consent
* Patient affiliated or beneficiary of a social security scheme

For alzheimer group : diagnosis of Alzheimer's disease according to NIA-AA 2024 criteria (presence of a pathogenic amyloid process in the cerebrospinal fluid)

For non alzheimer group : diagnosis of mild or major neurocognitive disorder according to Manuel diagnostique et statistique des troubles mentaux edition 5 (DSM-V) criteria, not linked to Alzheimer's disease (absence of pathogenic amyloid process in the cerebrospinal fluid)

Exclusion Criteria:

- Vulnerable people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial oxygen consumption of peripheral blood cells | At Baseline
  Comparison of the rate of mitochondrial oxygen consumption of peripheral blood cells between alzheimer (amyloid positive) and non-Alzheimer participant (amyloid negative) in pmol/min/cell mesured by Extracellular Flux Analyzer
Mitochondrial oxygen consumption of peripheral blood cells | At 1 year
  Comparison of the rate of mitochondrial oxygen consumption of peripheral blood cells between alzheimer (amyloid positive) and non-Alzheimer participant (amyloid negative) in pmol/min/cell mesured by Extracellular Flux Analyzer

SECONDARY OUTCOMES:
Mitochondrial metabolomic signature | At Baseline and at one year
  Description of the panel of mitochondrial metabolites of peripheral blood cells according to the status of the participants (amyloid positive vs amyloid negative).
Mini Mental State Examination Scores for Cognitive Impairment | At Baseline and at one year
  30 questions, good response to a question = 1, bad response to a question = 0, global scoring between 0 and 30,
  Pathological threshold according to the socio-cultural level :
  without diploma : total score <22 secondary education without the 3rd class : total score <23 secondary education from 3rd class to the senior year class (without bachelor degree) higher education : total score <26

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume SACCO, MD,PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, PACA, France

IPD SHARING:
Plan to Share IPD: No